CLINICAL TRIAL: NCT01398215
Title: Natural Orifice Translumenal Endoscopic Surgery (NOTES): Laparoscopic Assisted Transvaginal Ventral Hernia Repair
Acronym: NOTES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Garth Jacobsen, MD, Assistant Professor of Surgery, University of California, San Diego
Other Study IDs: 081038, 150520
Record Dates: First submitted 2011-07-14; First posted 2011-07-20 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Umbilical Hernia; Ventral Hernia
Keywords: umbilical hernia; ventral hernia
MeSH Terms: conditions — Hernia, Umbilical; Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- transvaginal NOTES
  Interventions: Procedure: transvaginal NOTES ventral hernia repair

INTERVENTIONS:
Procedure: transvaginal NOTES ventral hernia repair — ventral hernia repair via the transvaginal approach

SUMMARY:
This is a prospective chart review/data collection study of natural orifice translumenal endoscopic surgery (NOTES) for ventral hernia repair, that will include questionnaires administered throughout the study. Subjects enrolled will be those intending to have a transvaginal NOTES ventral hernia repair. Data will be collected and reviewed through 12 months post-op.

ELIGIBILITY:
Inclusion:

1. Umbilical or incisional hernia greater than 2 cm in size
2. Female, age 18-75
3. Mentally competent to give informed consent
4. Scheduled to undergo a transvaginal NOTES ventral hernia repair

Exclusion:

1. Pregnant women
2. Patients with defects measuring greater than 10 cm in size
3. Patients with complex hernias requiring fascial mobilization for closure
4. Morbidly obese patients (BMI >45)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who come to the UC San Diego Surgical Specialties clinic and have chosen to undergo a ventral hernia repair will be evaluated for participation in this tria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
To assess outcomes related to the transvaginal NOTES approach to laparoscopic ventral hernia repair (through data collection). | 1 Year
To assess pain associated with the transvaginal NOTES approach to laparoscopic ventral hernia repair (through data collection). | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Garth Jacobsen, M.D., Principal Investigator — UCSD
Locations (1):
- University of California, San Diego Medical Center, San Diego, California, United States